CLINICAL TRIAL: NCT02061605
Title: Phase-I Feasibility Trial To Study The Safety Of Laser Tissue Welding For Sealing Resected Kidney Surfaces After Laparoscopic Partial Nephrectomy
Brief Title: First-in-Human Safety Study Of Laser Tissue Welding For Surtureless Laparoscopic Partial Nephrectomy
Acronym: LTW-KIDNEY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Laser Tissue Welding, Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTW-LPN-01; R44DK094619-02 (NIH)
Record Dates: First submitted 2014-02-06; First posted 2014-02-13 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2019-02

CONDITIONS: Benign Renal Tumors; Malignant Renal Tumors
Keywords: Laparoscopic partial nephrectomy; Surgical hemostasis; Laser tissue welding; Tissue sealant
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser Tissue Welding Device (Experimental): The laser tissue welding device is intended for use in patients requiring laparoscopic surgery requiring hemostasis and sealing of the resected kidney after partial nephrectomy, and including those patients who are fully heparinized or have hemodilutional coagulation failure.
  The device's intended use is to seal the kidney surface using a laser to weld human albumin based biomaterials after surgical removal of kidney tumors during a laparoscopic partial nephrectomy.
  Interventions: Device: Laser Tissue Welding Device

INTERVENTIONS:
Device: Laser Tissue Welding Device — Laparoscopic partial nephrectomy will be robotically assisted using the second generation da Vinci® Surgical System. Once the tumor is resected with laparoscopic scissors with a margin of healthy tissue, the solder will be dripped onto the cut surface of the parenchyma. A laparoscopic rigid 5mm spot-size laser hand-piece will be passed through the 10-mm port. The diode laser will be then used to weld a thin layer of solder onto the cut parenchymal surface. The 60 Watt 810-nm diode laser will be set to deliver continuous energy. During soldering, the tip of the laparoscopic laser hand-piece will be maintained 1 to 2 cm from the renal surface to generate a spot size of approximately 5 mm. Each spot will be treated with the laser until the color of the solder changes from green to white. The renal pedicle clamp will be removed to allow renal blood supply to be restored and the surgical site inspected for evidence of bleeding for 10 minutes prior to completing the surgical procedure.

SUMMARY:
The objective of this pilot study will be to obtain a clinical safety and efficacy endpoint profile of laser tissue welding therapy for sealing the resected kidney surface after laparoscopic partial nephrectomy required for removal of resectable benign or malignant renal tumors in 10 patients.

DETAILED DESCRIPTION:
SCIENTIFIC RATIONALE:

The use of partial nephrectomy to treat small newly diagnosed kidney tumors is vastly under-used as per NCI statistics (http://www.cancer.gov/cancertopics/treatment/partial-nephrectomy0208).

As per the Surveillance, Epidemiology and End Results (SEER) Program, (http://seer.cancer.gov/statfacts/html/kidrp.html), the prevalence of cancer of the kidney and renal pelvis is 296,074 while the estimated new cases are 46,410 and deaths 13,040 in the United States in 2010 (www.cancer.gov/cancertopics/types/kidney).

There has been an increase in detection of incidental small renal mass (≤ 4cm) cases (TNM staging T1a) due to widespread use of ultrasound and abdominal cross sectional imaging (CT, MRI) and thus an increase in the amount of renal surgery performed. Current surgical practice for nephron sparing surgery allows at least 1 cm margin of normal tissue around the tumor3. This is the stage when curative resections are possible.

During a partial nephrectomy, the renal artery is clamped to minimize bleeding while resecting the tumor. Since a major reconstruction is required with suturing, clamp time can be significant, anywhere between 15 and 45 minutes. It has been repeatedly shown that reducing clamp time preserves renal function and that there is significant damage to the kidney if the renal artery is clamped for more than 30 minutes. This is especially crucial when dealing with patients with hypertension, diabetes, chronic renal failure or a tumor in a single kidney. Extended clamp time can result in decreased renal function and ultimately the need for dialysis at some point. Because of the inherent difficulties of laparoscopic suturing, this has not been widely used particularly in view of the risk of prolonged warm ischemia time. Many patients therefore undergo a radical nephrectomy instead of a nephron sparing procedure. Hemorrhage 9.5% (1) , is the major complication following partial nephrectomy. Besides bleeding (1) urinary fistula (4.5%), ureteral obstruction, and renal insufficiency due to prolonged warm ischemia times are further complications of partial nephrectomy.

Laser Tissue Welding is the first combination (laser and biologic) class III surgical device intended to join and seal tissues accurately and instantly. The treatment process uses thermal energy created when a laser excites photosensitive dye molecules, to coagulate the protein albumin which transforms from a liquid to a solid instantly. Laser tissue welding creates a non-compressive, non-ablative sealing of tissues with microscopic thermal damage. This combination of a laser with albumin biologics stops bleeding and fluid leaks in nanoseconds without using sutures, hemostatic clotting factors (platelets/thrombin/fibrin), thermal or cryoablation. (Video: http://www.lasertissuewelding.com/application.aspx?AID=8)

ELIGIBILITY:
Inclusion Criteria:

1. T1a (< 4 cm). All resectable benign, primary or secondary malignant tumors of one kidney. No bi-lateral disease.
2. Serum creatinine: ≤ 2.5 mg/dL
3. Glomerular filtration rate greater than ≥ 50 ml/min/m2
4. Platelet count ≥ 50,000/mm3
5. Prothrombin time < 18 seconds
6. Partial thromboplastin time (PTT) ≤ 1.5 times control
7. Serum albumin levels > 3g/dL (Normal range 3.5 to 5 g/dL)

Exclusion Criteria:

1. Age younger than 18 years old
2. Severe uncorrected hypertension
3. Uncorrectable coagulopathies
4. Pregnancy
5. Active urinary tract infection
6. T1b (>4 cm) lesion and above
7. Systemic or local infection
8. Subject has known allergy or intolerance to iodine or human serum albumin
9. Recent febrile illness that precludes or delays participation pre-operatively
10. Treatment with another investigational drug or other intervention during the study and follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Operative Blood Loss | Day 1
  Operative blood loss is defined by: Volume of blood in the suction bottles, volume of blood clots, and weight of surgical towels before and after use.
  Clinical assessment of the blood loss: Clinical drop in hemoglobin (1 gm. % = 300 ml) without hemo-dilution. Therefore is correlated with blood products transfused to compensate for the blood lost during surgery.
Postoperative Blood Loss | Up to 30 days
  Clinical assessment of the blood loss:
  1. Clinical drop in hemoglobin (1 gm. % = 300 ml) without hemodilution. Therefore is correlated with blood products transfused to compensate for the blood lost post-operatively.
  2. Correlated to post-operative JP tube drainage, amount and type.

SECONDARY OUTCOMES:
Secondary hemorrhage or hematoma (safety issue no. 1) | Up to 12 months
  Post-operative blood loss requiring return to the operating room
Post-operative urinary leakage/ urinoma (safety issue no. 2) | Up to 12 months
  Urinary leakage is measured in drainage bottles (ml/day) following surgery till a drain placed during the operation is removed before patient discharge. Accumulation of fluids around the kidney (blood or urine) will be assessed with U/S and CT scan at the mentioned time points.
Secondary infection, intra-abdominal abscess formation and septicemia (safety issue no. 3) | Up to 12 months
  Surgical space abscess
Urinary stone formation (safety issue no. 4) | Up to 12 months
  To see if the protein solder is a nidus for stone formation

OTHER OUTCOMES:
Total operating time (minutes) (Duration Metric -1) | Day 1
  Observed operative period
Nephrectomy clamp time (minutes) (Duration Metric-2) | Day 1
  Observed intra-operatively. Assesses organ ischemia time and will correlate with compromised renal function post-surgery.
Laser tissue welding time (sec/cm2) (Duration Metric-3) | Day 1
  Observed intra-operatively:
  Cumulative time to complete hemostasis. This will be compared to current standard of care time-to-hemostasis using suture closure which is anywhere between 15 and 45 minutes since a major renal reconstruction is required with suturing and therefore correlated to significant clamp time, renal ischemia and renal dysfunction.
Length of ICU stay (Duration Metric-4) | Up to 12 months
  Number of days spent in intensive care unit (ICU).
Length hospital stay ((Duration Metric-5) | Up to 12 months
  Total time spent as an in-patient

CONTACTS AND LOCATIONS:
Overall Officials: RICHARD LINK, M.D., Principal Investigator — Department of Urology, Baylor College of Medicine
Locations (1):
- St. Luke's Episcopal Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Laser Tissue Welding, Inc — http://www.lasertissuewelding.com/